CLINICAL TRIAL: NCT06034314
Title: Investigation of the Effects of Cannabis on the Immune-genome in People With HIV
Brief Title: Oral Dronabinol-HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000035807; 1R01DA052846-01 (NIH)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HIV
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- People with HIV (PWH) with Cannabis use (Experimental): PWH with cannabis use
  Interventions: Drug: Dronabinol Capsules
- People without HIV (PWoH) with Cannabis use (Experimental): PWoH with Cannabis use
  Interventions: Drug: Dronabinol Capsules

INTERVENTIONS:
Drug: Dronabinol Capsules — Two 10 mg Dronabinol capsules will be administered orally, for a total of 20mg, on test day.
  Other Names: Marinol; Syndros

SUMMARY:
The purpose of this study is to define the mechanisms of cannabis on the genome of people with HIV who use cannabis. The investigator aims to better understand the effect of Dronabinol on immune and inflammatory functions, and whether these changes are HIV-status dependent. This research may better inform public health policy regarding cannabis use. Depending on the results, additional studies may also build upon this research to develop more effective and specific treatments for cannabis use associated disorders.

ELIGIBILITY:
PWH Inclusion Criteria:

* Current or past Cannabis use.
* HIV-positive on antiretroviral therapy.
* Meet criteria of viral suppression (viral load less than approximately 400 copies/ml).
* Good physical and mental health as determined by history, the SCID, collateral information, physical and laboratory examinations, ECG, and vital signs.
* Women of Childbearing Potential: Must agree to use or have their partner use one acceptable method of birth control throughout the study, at the discretion of the principal investigator.

PWoH Inclusion Criteria:

* Current or past Cannabis use.
* Good physical and mental health as determined by history, the SCID, collateral information, physical and laboratory examinations, ECG, and vital signs.
* Women of Childbearing Potential: Must agree to use or have their partner use one acceptable method of birth control throughout the study, at the discretion of the principal investigator.

Exclusion Criteria:

* Cannabis naïve individuals.
* Under the age of 18 years.
* Unable to provide written informed consent.
* Unable to read or write in English.
* Unable to tolerate the effects of smoking approximately half a joint of cannabis (or equivalent), at the discretion of the principal investigator.
* Major or clinically unstable medical conditions (e.g., myocardial infarction, hypertension, clinically significant head injury or loss of consciousness).
* IQ less than 80.
* Diagnosis of psychosis confirmed by SCID.
* Other medical, psychiatric, or psychosocial history that is deemed unsuitable for participation in study per PI.
* Has donated blood within the last 8 weeks.
* Sesame oil allergy.
* Concomitant use of other drugs that cause dizziness, confusion, sedation, or somnolence such as CNS depressants (e.g., barbiturates, benzodiazepines, ethanol, lithium, opioids, buspirone, scopolamine, antihistamines, tricyclic antidepressants, other anticholinergic agents, muscle relaxants).
* Patients with cardiac disorders or concomitant use of other drugs that are associated with similar cardiac effects (e.g., amphetamines, other sympathomimetic agents, atropine, amoxapine, scopolamine, antihistamines, other anticholinergic agents, amitriptyline, desipramine, other tricyclic antidepressants).
* Patients with a history of seizures, including those receiving anti-epileptic medication or with other factors that can lower the seizure threshold.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dronabinol-induced transcriptome profile in blood using single cell (sc)RNA-seq | Baseline, 120 minutes post-Dronabinol and 360 minutes post-Dronabinol
  Changes at baseline, 120 minutes, and 360 minutes post oral Dronabinol. Transcriptome will be profiled by using single cell (sc)RNA-seq in blood samples. A panel of 45 cytokines and profiling of 37 immune cell types will be assessed for functional evaluation after Dronabinol administration.

SECONDARY OUTCOMES:
Change in Dronabinol-induced chromatin structure profile in blood samples using single cell (sc)ATAC-seq | Baseline, 120 minutes post-Dronabinol and 360 minutes post-Dronabinol, up 5 years
  Changes in chromatin structure will be profiled by using (sc)ATAC-seq and capture methylome sequencing in a subset of samples from the primary outcome. The investigator expects to identify the differentially accessible regions and DNA methylation regions between pre- and post-Dronabinol administration that are correlated with Dronabinol-induced immune gene expression in each cell type.
Identification of Dronabinol related cellular gene networks in blood samples | up 5 years
  Data from scRNA-seq (Outcome 1) and scATAC-seq (Outcome 2) will be used to establish a computational strategy to identify cell type specific gene networks for Dronabinol response in PWoH and PWH samples separately and by HIV status.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Xu, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No